CLINICAL TRIAL: NCT07049666
Title: Effects of Preoxygenation With Bag-valve-mask and Noninvasive Mechanical Ventilation on Oxygenation and Hemodynamics: A Randomized Controlled Study
Brief Title: Preoxygenation and Hemodynamics With Bag-valve-mask and Noninvasive Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KA22/426
Record Dates: First submitted 2025-06-17; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Preoxygenation
Keywords: Preoxygenation; bag-valve-mask; noninvasive mechanical ventilation; hemodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bag-valve mask ventilation (Experimental): Preoxygenation was administered utilizing a Compower (Fujian, China) BVM equipped with an oxygen reservoir, coupled with a correctly fitted oronasal mask. This preoxygenation procedure spanned three minutes, with an oxygen flow rate set at 15 liters per minute.
  Interventions: Device: Bag-valve mask; Device: Noninvasive mechanical ventilation
- noninvasive mechanical ventilation (Active Comparator): Preoxygenation was conducted over a three-minute period using NIMV employing a properly fitted oronasal mask. This was facilitated by the Servo S (Maquet, Solna, Sweden) mechanical ventilator operating in pressure support mode. The preoxygenation protocol entailed the administration of 100% FiO2, applying Positive End-Expiratory Pressure (PEEP) set at 5 cmH2O, delivering breaths at a frequency of 15 per minute, and providing a tidal volume ranging between 6 to 8 ml/kg of body weight.
  Interventions: Device: Bag-valve mask; Device: Noninvasive mechanical ventilation

INTERVENTIONS:
Device: Bag-valve mask — A BVM equipped with an oxygen reservoir, coupled with a correctly fitted oronasal mask was used.
Device: Noninvasive mechanical ventilation — Preoxygenation was conducted over a three-minute period using NIMV employing a properly fitted oronasal mask. This was facilitated by a mechanical ventilator operating in pressure support mode. The preoxygenation protocol entailed the administration of 100% FiO2, applying Positive End-Expiratory Pressure set at 5 cmH2O, delivering breaths at a frequency of 15 per minute, and providing a tidal volume ranging between 6 to 8 ml/kg of body weight.

SUMMARY:
Hypoxemia refers to low blood oxygen levels, while hypoxia denotes low tissue oxygen levels. Both conditions pose life-threatening risks when precautions are not adequately taken or when risks are not effectively managed. Intubation represents a critical phase that can lead to a decrease in arterial oxyhemoglobin levels. Two frequently employed techniques for preoxygenation and ventilation during intubation are bag-valve mask (BVM) ventilation and noninvasive mechanical ventilation (NIMV). The aim of this study was to evaluate the efficacy and safety of BMV and the NIMV.

DETAILED DESCRIPTION:
Ventilation and intubation challenges increase the risk of arterial desaturation, emphasizing the importance of careful management during this process. Throughout the intubation process, the oxygen reserves within the lung, plasma, hemoglobin, body mass index (BMI) play a critical role in meeting the tissue oxygen demand. Preoxygenation serves to extend the time window for intubation safely. The quantity of available oxygen reserve and the duration of the apneic period represent the primary determinants for the occurrence of hypoxemia during intubation.

Anticipating difficult intubation is crucial, as it often prolongs both the duration of intubation and the apneic period. The Intubation Difficulty Scale (IDS) is commonly utilized to predict the likelihood of encountering difficult intubation scenarios. It is imperative to select the appropriate preoxygenation technique, particularly in patients with a high IDS, to mitigate the risk of desaturation during the intubation process.

Two frequently employed techniques for preoxygenation and ventilation during intubation are BVM ventilation and NIMV. Preoxygenation, also referred to as denitrogenation, has the potential to induce atelectasis. However, this complication can be mitigated with positive pressure ventilation (PPV), which not only aids in maintaining oxygen levels but also exerts effects on the circulatory system. Hypotension is the most common symptom that occurs as a result of the interaction of the respiratory and circulatory systems.

The objective of this study was to evaluate and compare the impacts of preoxygenation with BVM and NIMV techniques on oxygenation and hemodynamic parameters specifically during the apneic period of endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Having a partial arterial oxygen pressure (PaO2)/fraction of inspired oxygen (FiO2) ratio exceeding 200
* Consented to participate

Exclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) Physical Status Classification System Score 4
* Patients with a Mallampati Score greater than 3
* Patients with a history of difficult intubation
* Patients who are pregnancy
* Patients who have hypoxia (defined as a PaO2/FiO2 ratio less than 200)
* Patients with heart failure
* Patients with chronic obstructive pulmonary disease
* Patients who undergoing emergency surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2022-12-26 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in partial pressure of oxygen in arterial blood (PaO₂) values after 3 minutes of preoxygenation | At the end of 3 minutes of preoxygenation
  To compare PaO₂ between study groups after 3 minutes of preoxygenation (Unit of Measure: mmHg)
Change in partial pressure of carbon dioxide in arterial blood (PaCO₂) values after 3 minutes of preoxygenation | At the end of 3 minutes of preoxygenation
  To compare PaCO₂ between study groups after 3 minutes of preoxygenation (Unit of Measure: mmHg)

SECONDARY OUTCOMES:
Change in systolic blood pressure | At the 5th minute after intubation
  Systolic arterial pressure will be recorded and compared between groups at the 5th minute after intubation
Change in diastolic blood pressure | At the 5th minute after intubation
  Diastolic arterial pressure will be recorded and compared between groups. (Unit of Measure: mmHg)
Change in mean arterial pressure (MAP) | At the 5th minute after intubation
  MAP will be recorded at the 5th minute after intubation (Unit of Measure: mmHg)
Change in heart rate | At the 5th minute after intubation
  Heart rate will be monitored and compared between groups at the 5th minute after intubation. [Unit of Measure: beats per minute (bpm)]
Change in peripheral oxygen saturation (SpO₂) | At the 5th minute after intubation
  SpO₂ will be monitored continuously and analyzed at the 5th minute after intubation. (Unit of Measure: percentage (%))

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Adana, Yuregır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321